CLINICAL TRIAL: NCT07095985
Title: A Retrospective Cohort Study Evaluating the Safety and Clinical Efficacy of a Novel Anastomotic Technique for Restoring Ileocecal Valve Function During Laparoscopic Radical Resection of Right-Sided Colon Cancer
Brief Title: Novel Ileocecal Valve-Sparing Anastomosis in Laparoscopic Right Hemicolectomy
Status: Completed | Type: Observational
Sponsor: Army Medical University, China (Other)
Responsible Party: Principal Investigator, Weidong Xiao, Head of General Surgery, Clinical Professor, Army Medical University, China
Other Study IDs: RISE anastomosis 001
Record Dates: First submitted 2025-06-26; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Radical Right Hemicolectomy
Keywords: Right hemicolectomy; Ileocecal valve reconstruction; RISE anastomosis; Laparoscopic surgery; Colon cancer; Anastomotic technique; Bowel function; Retrospective cohort study
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RISE anastomosis: Following right hemicolectomy, the novel RISE-ICVR technique involves everting the ileal stump to create an artificial valve, implanting it into a colonic wall incision, and securing it with circumferential sutures.
- Conventional Anastomosis Group: In contrast, the conventional approach uses a linear stapler to perform a side-to-side ileocolic anastomosis.

SUMMARY:
This is a single-center retrospective cohort study conducted by the Department of General Surgery at the Second Affiliated Hospital of Army Medical University (Xinqiao Hospital). The study aims to evaluate the safety and clinical efficacy of a novel anastomotic technique designed to reconstruct ileocecal valve (ICV) function during laparoscopic right hemicolectomy for right-sided colon cancer.

Background: Standard right hemicolectomy necessitates resection of the ICV, a critical structure regulating ileocolonic transit and acting as a bacterial barrier. Its loss can lead to small intestinal bacterial overgrowth (SIBO), diarrhea, malabsorption, and reduced quality of life. While preserving the ICV is ideal when oncologically feasible, it's often unavoidable. This study proposes an innovative anastomosis technique ("Revolute Insert Side-End Ileocecal Valve Reconstruction" - "RISE anastomosis") to functionally reconstruct the ICV.

Study Design:

Population: 50 patients who underwent laparoscopic right hemicolectomy at the center, meeting inclusion/exclusion criteria (age 18-80, ASA ≤3, primary tumors in appendix, cecum, ascending colon, hepatic flexure, or proximal 1/3 transverse colon, complete data).

Groups:

Conventional Anastomosis Group (n=30): Standard side-to-side ileocolic anastomosis using a linear stapler.

RISE anastomosis Group (n=20): Novel technique involving everting the ileal stump with sutures to create an artificial valve, then implanting it into an incision on the colonic wall and suturing it circumferentially.

Primary Objective: Assess safety and feasibility of RISE anastomosis.

Secondary Objective: Evaluate the clinical efficacy of RISE anastomosis on bowel function recovery.

Key Outcomes:

Safety (Primary): 30-day postoperative complications (anastomotic leak, bleeding, stricture), severe complications (Clavien-Dindo).

Efficacy (Secondary): Time to first flatus, first defecation, first formed stool; Bristol stool scale; defecation frequency/urgency; incontinence rates; length of stay; reoperation/readmission rates.

Other: Operative time, anastomosis time, blood loss, lymph node yield, inflammatory markers, follow-up assessments (contrast studies, endoscopy).

Data Analysis: Data extracted from electronic medical records. Statistical analysis using SPSS 22.0 (χ² test for categorical data, t-test for normally distributed continuous data; significance p<0.05).

Ethics: Approved by the institutional ethics committee. Conducted in accordance with the Declaration of Helsinki and Chinese regulations. Patient privacy and data confidentiality are prioritized.

Timeline: Patient data collection and analysis (Jun-Aug 2024); Statistical analysis and manuscript preparation (Sep-Dec 2024).

Significance: This study investigates a potentially transformative surgical technique. If proven safe and effective, RISE anastomosis could significantly improve postoperative bowel function and quality of life for patients requiring ICV resection during right hemicolectomy, addressing a major unmet clinical need related to ICV loss.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification of II-III.
* Patients newly diagnosed with tumors located in the appendix, ileocecal region, ascending colon, hepatic flexure, or the right one-third of the transverse colon, or those scheduled to undergo laparoscopic right hemicolectomy.
* No history of other gastrointestinal diseases (excluding intestinal polyps and gallstones).
* Willingness to participate in the study with signed informed consent.
* Complete clinical data available.

Exclusion Criteria:

* Presence of malignancies in other anatomical sites.
* Tumor invasion into adjacent organs.
* Presence of infectious or autoimmune diseases (e.g., Crohn's disease).
* Congenital or acquired metabolic disorders.
* Use of antibiotics or other microbiota-altering medications within one month before enrollment.
* Changes in surgical plan such that the resection does not include the ileocecal valve.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who visited Xinqiao Hospital and were diagnosed with right-sided colon cancer
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
30-day postoperative complications (anastomotic leak, bleeding, stricture), severe complications (Clavien-Dindo). | from day1 to day30 after surgery
  After the surgery, continuously record whether the patient has any adverse reactions until 30 days postoperatively, and score the severity of the adverse reactions according to the Clavien-Dindo classification.

SECONDARY OUTCOMES:
Time to first flatus | from day1 to day7 after surgery
  Record the time of the patient's first bowel movement after surgery.
Time to first formed stool | from day1 to day30 after surgery
  Record the time of the patient's first formed stool after surgery.

OTHER OUTCOMES:
Operative time | During the operation
  Surgical time, as recorded on the anesthesia record.
Anastomosis time | During the operation
  Anastomosis time: Calculated based on the surgical video recordings.
Blood loss | During the operation
  blood loss, as recorded on the anesthesia record.
Inflammatory markers | from day1 to day7 after surgery
  The value of white blood cell count in the complete blood count (CBC) test.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Xiao, MD, Study Chair — Second Affiliated Hospital of Army Medical University
Locations (1):
- Xinqiao Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
We are currently planning to conduct a series of studies. As data sharing will be postponed until all studies have been completed, the data will not be made available at this time.

DOCUMENTS (1):
  • Study Protocol (2025-06-26): https://cdn.clinicaltrials.gov/large-docs/85/NCT07095985/Prot_000.pdf